CLINICAL TRIAL: NCT01659008
Title: Estradiol Versus Tranexamic Acid on the Amount and Duration of Acute Cyclic Heavy Menstrual Bleeding
Brief Title: Estradiol vs Lysteda in Treatment of Heavy Menstrual Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kay I Waud MD PhD (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Sponsor-Investigator, Kay I Waud MD PhD, principal investigator, FELLOW physician PGY6, Eastern Virginia Medical School
Organization: Eastern Virginia Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-01-FB-0003
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Menstrual Cycle and Uterine Bleeding Disorders
Keywords: acute cyclical heavy menstrual bleeding
MeSH Terms: interventions — Estradiol; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- estradiol (Experimental): estradiol PO 0.5mg 2 tabs three times a day for 2 days
  Interventions: Drug: Estradiol
- Lysteda (Experimental): Lysteda 650mg PO 2 tabs three times a day for 2 days
  Interventions: Drug: Lysteda

INTERVENTIONS:
Drug: Estradiol
  Arms: estradiol
Drug: Lysteda
  Arms: Lysteda

SUMMARY:
Treatment with Estradiol is non-inferior to treatment with Tranexamic acid in reducing the amount and duration of menstrual blood loss in women with cyclic heavy menstrual bleeding

DETAILED DESCRIPTION:
BACKGROUND: The acute onset of Heavy Menstrual Bleeding (HMB) during menses results in women seeking care in the Emergency Department. The current management of HMB among our residents uses combination oral contraceptives or oral progestins. The residents in the Emergency Department often send women home without any therapeutic intervention. There is no Regulatory Agency approved therapy for acute HMB. The etiology of HMB is not well understood. Two potential causes are changes in endometrial prostaglandins and increased fibrinolytic activity in the endometrium.

Specific Aim 1 is to investigate and compare the effect of oral estradiol compared to tranexamic acid in reducing blood loss and the duration of bleeding during an acute episode HMB.

Specific Aim 2 is to evaluate the effect of estradiol and tranexamic acid on possible causes of the acute HMB by measuring prostaglandins and Plasminogen activator in menstrual effluent at the end of treatment.

METHODS: This is a randomized, double-blind, controlled, parallel-group, non-inferiority trial, with participants between the ages 18 and 45 years, with acute cyclic heavy menstrual bleeding enrolled during an emergency room visit. Participants are randomized to receive 48 hours' treatment with 1.3 mg oral tranexamic acid or 1.0 mg oral estradiol three times a day. The primary endpoint is reduction in the amount of menstrual effluent. Sample size was calculated based on detecting less than 30 ml difference between the mean menstrual blood loss of the two treatment groups. Amount of blood loss is quantified by alkaline hematin method on extraction of menstrual pads and tampons. Secondary outcome is the variation of hemostatic factors in the menstrual effluent in two treatment groups by collecting menstrual effluent and quantitating prostaglandins, Plasminogen activators, Plasminogen activator inhibitors, and vascular endothelial growth factor.

ANTICIPATED OUTCOMES: The investigators anticipate a reduction in mean menstrual blood loss in both treatment groups. Compared with participants treated with estradiol, the group treated with tranexamic acid will not have statistically significant change in reduction of menstrual effluent. We also anticipate changes in different local hemostatic factors in menstrual effluent specific to the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18-45 years old
* Hemoglobin concentration: less than or equal to 11.5 g/dL, greater than or equal to 8.0 g/dL
* BMI: less than or equal to 35
* Menstrual cycle: previous menstrual cycle interval between 26 to 34 days with less than or equal to 10 days of bleeding
* Contraception: at least two months from implant removal, or six months from their last depo-provera or depo-Lupron injection, or recently(at least 2 months) discontinued oral, patch or intravaginal ring contraceptives
* On cycle day 1-3 of the current menstrual bleeding episode

Exclusion Criteria:

* NSAID, or aspirin containing medications during the 48 hours preceding the current ER visit
* Estrogen or progestin treatment during the 30 days preceding the current ER visit
* Using Paraguard
* Pregnant and or lactating
* History of endometrial ablation
* Women with thromboembolic disease, or coagulopathy
* Women with history of myocardial infarction, or cerebrovascular occlusion
* Uncontrolled high blood pressure (blood pressure greater than 150/90)
* Sensitivity to estrogen, or tranexamic acid

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
menstrual blood loss | 48 hours
  reduction in mean menstrual blood loss in both treatment groups

SECONDARY OUTCOMES:
changes in local hemostatic factors | 48 hours
  changes in local, endometrial hemostatic factors in both treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Kay I Waud, MD PhD, Principal Investigator — Eastern Virginia Medical School department of obstetrics and gynecology
Locations (2):
- United States (2):
  - Jones Institue Clinical Research Center, Norfolk, Virginia
  - Sentara Norfolk General Emergency Department, Norfolk, Virginia